CLINICAL TRIAL: NCT07213011
Title: Effects of Neck Static Stretching and Self-myofascial Release on Local and Remote Range of Motion: a Randomized Crossover Trial
Brief Title: Effects of Static Stretching and Self-myofascial Release on Local and Remote Range of Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Ewan Thomas, Associate Professor in the Department of Psychology, Education Sciences and Human Movement, University of Palermo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RE 306/2025
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Health; Healthy Participants; Healthy Subjects; Healthy Young People; Healthy Young Adults; Stretching; Myofascial Release; Massage Effect
Keywords: stretch; massage roller; cervical; mobility; remote effects

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Static stretching (Experimental): The neck static stretching protocol consisted of four sets of 45 seconds each, with 45-second rest intervals between sets, resulting in a total intervention time of three minutes. Participants remained seated in an upright position and executed the stretch by gently inclining the head in an anterolateral direction, forward and to the left, while using the contralateral (left) hand to assist the movement. This positioning was intended to specifically target and elongate the right posterolateral neck musculature.
  Interventions: Other: Neck static stretching
- Self-myofascial release (Experimental): For the neck self-myofascial release intervention, a Theraband® Roller Massager (The Hygenic Corporation, Akron, OH, USA) was utilized. This device features a rigid plastic core encased in high-density foam with a grooved surface, designed to facilitate both superficial and deeper tissue stimulation. The self-myofascial release protocol consisted of four sets, each comprising 45 rhythmic rolling movements performed at a standardized cadence of one roll per second, totaling three minutes of intervention time. The rolling tempo was regulated using a metronome application (Tempo Lite, version 5.0.8; Apple App Store). A 45-second rest interval was provided between sets. While seated, participants self-administered the rolling technique to the right posterolateral region of the neck, ensuring coverage of the largest possible surface area. To optimize tissue elongation, the head was maintained in a gently inclined anterolateral position, forward and to the left, throughout the intervention.
  Interventions: Other: Neck self-myofascial release
- Control (No Intervention): In the control condition (CC), participants remained seated quietly on a chair for a period of 6 minutes, matching the duration of the static stretching and self-myofascial release protocols, but without performing any active intervention, between the baseline and post assessments.

INTERVENTIONS:
Other: Neck static stretching — The neck static stretching (SS) protocol consisted of four sets, each lasting 45 seconds, interspersed with 45-second recovery periods (total intervention time: 3 minutes). While seated on a chair, participants performed the stretch by gently inclining the head forward and to the left in an antero-lateral direction and assisting the movement with the contralateral (left) hand to specifically elongate the right posterolateral neck region.
  Arms: Static stretching
Other: Neck self-myofascial release — For the self-myofascial release (SMR) intervention, a Theraband® roller massager was employed. The device consists of a rigid plastic core surrounded by dense foam, designed with a grooved surface to facilitate both superficial and deeper tissue stimulation. The SMR protocol comprised four sets (total intervention time: 3 minutes), during which participants executed 45 rhythmic rolling movements per set at a cadence of one roll per second. The tempo was standardized using a metronome application. For the SMR condition, the protocol included 45-second recovery intervals between sets. Participants, seated on a chair, were instructed to perform self-administered rolling on the right posterolateral neck region using the massage roller and to cover the largest possible area of the posterolateral neck region during the rolling, with the head gently inclined forward and to the left in an antero-lateral direction.
  Arms: Self-myofascial release

SUMMARY:
Static stretching and self-myofascial release are commonly used techniques to improve joint mobility, primarily through mechanisms such as reduced tissue stiffness, increased stretch tolerance, and warming effects. Emerging evidence suggests that these interventions may also elicit remote effects, improving range of motion in body segments distant from the site of application. These non-local adaptations are thought to occur via mechanisms such as myofascial force transmission, systemic increases in stretch tolerance, or global neuromuscular responses. This phenomenon may have important clinical implications, particularly in scenarios where direct treatment of a target area is limited due to pain, injury, or immobilization.

Therefore, this study explores the potential for local and remote effects of static stretching and self-myofascial release applied to the right posterolateral neck region. Specifically, this study investigates whether targeted cervical interventions can acutely improve not only cervical range of motion but also hip flexion range of motion on the ipsilateral (right) side. The proposed mechanisms include reductions in tissue stiffness, increased stretch tolerance and pressure pain threshold, and the transmission of mechanical forces along myofascial chains, particularly the "superficial back line," which anatomically connects the cervical region to the posterior lower limb. The primary aim of this study was to compare the acute effects of neck static stretching and neck self-myofascial release using a massage roller on both local (cervical) and remote (right hip) ROM.

DETAILED DESCRIPTION:
All outcome data will be expressed as mean ± standard deviation. The reliability of baseline measurements (T0) will be assessed using intraclass correlation coefficients (ICC) for all variables. After verifying the distribution of the data, potential baseline differences among the three experimental conditions will be assessed (stretching, myofascial release, and control) through a one-way analysis of variance (ANOVA).

To examine differences in the main outcomes, a repeated-measures ANOVA (3 conditions × 2 time points) will be conducted. When a significant condition × time interaction is detected, post hoc analyses with Scheffé corrections will be applied to determine specific between and within-group differences. Effect sizes will be reported as partial eta squared (η²p). Statistical significance will be set at p < 0.05 for all analyses

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants aged 18 or older.

Exclusion Criteria:

* orthopedic or neurological disorders;
* current and recent injuries or damage to the upper and lower limbs.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-05-14 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Range Of Motion | During each condition (SS, SMR, CC), hip and cervical ROM was collected at two time-points: upon arrival (T0) and immediately following the assigned condition (T1).
  Right hip flexion range of motion (ROM) was assessed using the Active Straight Leg Raise test. Participants lay in a supine position with the test knee fully extended and the ankle dorsiflexed, a setup intended to specifically assess hamstring extensibility. Hip flexion was measured in degrees using the GYKO inertial measurement unit.
  Cervical ROM was evaluated with participants seated and secured to the chair at the chest level using inelastic straps to limit trunk movement. The GYKO accelerometer was positioned on the forehead via a head strap and recorded active cervical movements in flexion, extension, right and left rotation, and right and left inclination.
  The investigators collected three ROM measurements for each movement (hip flexion, cervical flexion/extension, right and left cervical rotation, right and left cervical inclination) and for each time point (T0 and T1), then used the average of the three measurements for statistical analysis.
Tissue Hardness | During each condition (SS, SMR, CC), cervical and hamstring TH was collected at two time-points: upon arrival (T0) and immediately following the assigned condition (T1).
  Tissue hardness (TH) nwas assessed using a portable TH meter (NEUTONE TDM-N1; TRY-ALL Corp., Chiba, Japan). For cervical TH assessment, the spinous process of C7 served as the anatomical landmark. Measurements were taken at two locations, positioned 2 cm lateral to the right and left of the C7 spinous process. Assessment of TH in the right knee flexors was conducted using the ischial tuberosity as the proximal reference point and the popliteal fossa as the distal landmark. Measurements were obtained at two specific sites located in the proximal third of the posterior thigh: a lateral site corresponding to the biceps femoris and a medial site corresponding to the semitendinosus/semimembranosus muscle complex. All TH measurements were performed with participants in a prone position on a medical examination bed. Participants were instructed to remain relaxed throughout the procedure. For each time point (T0 and T1), three consecutive measurements were taken per anatomical site.
Pain Pressure Threshold | During each condition (SS, SMR, CC), cervical and hamstring PPT was collected at two time-points: upon arrival (T0) and immediately following the assigned condition (T1).
  Pain pressure threshold (PPT) was measured using a portable digital algometer (FPX 25 Pain Tester, Wagner Instruments, CT, USA). Participant positioning and the anatomical testing sites were identical to those used for the TH assessments. The algometer probe was applied perpendicularly to the muscle fibers, and pressure was manually increased at a constant rate of 1 kg·s-¹ by the same trained investigator to ensure consistency. Participants were instructed to verbally indicate "stop" at the point where the sensation first transitioned from pressure to pain. The corresponding value displayed on the algometer at that moment, expressed in kg·cm-², was recorded as the PPT. The investigators collected three PPT measurements for each anatomical site and time point (T0 and T1), then used the average of the three measurements for statistical analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Palermo, Palermo, Italy